CLINICAL TRIAL: NCT00395746
Title: Effect of Liraglutide in Combination With Sulfonylurea (SU) on Glycaemic Control in Subjects With Type 2 Diabetes
Brief Title: Effect of Liraglutide in Combination With Sulfonylurea (SU) on Blood Glucose Control in Subjects With Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN2211-1701; JapicCTI-060324 (Registry Identifier: japic)
Record Dates: First submitted 2006-11-02; First posted 2006-11-03 (Estimated); Results first posted 2010-03-12 (Estimated); Last update posted 2017-03-08 (Actual); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Sulfonylurea Compounds; Liraglutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 0.6 mg + SU (Experimental): Liraglutide 0.6 mg + sulphonylurea
  Interventions: Drug: sulfonylurea; Drug: liraglutide
- 0.9 mg + SU (Experimental): Liraglutide 0.9 mg + sulphonylurea
  Interventions: Drug: sulfonylurea; Drug: liraglutide
- SU Mono - 1 (Placebo Comparator): Liraglutide placebo 0.6 mg + sulphonylurea
  Interventions: Drug: sulfonylurea
- SU Mono - 2 (Placebo Comparator): Liraglutide placebo 0.9 mg + sulphonylurea
  Interventions: Drug: sulfonylurea

INTERVENTIONS:
Drug: sulfonylurea — SU agent
Drug: liraglutide — Liraglutide 0.6 mg/day or placebo. Injected s.c. (under the skin) once daily.
  Arms: 0.6 mg + SU
Drug: liraglutide — Liraglutide 0.9 mg/day or placebo. Injected s.c. (under the skin) once daily.
  Arms: 0.9 mg + SU

SUMMARY:
This trial is conducted in Japan. The trial aims for comparison of the effect on glycaemic control of liraglutide in combination with sulphonylurea agent (SU) compared to SU monotherapy, as assessed by HbA1c after 24 weeks and 52 weeks in subjects with type 2 diabetes. Liraglutide will be compared to placebo, in combination with SU. Trial has a randomisation period of 24 weeks followed by a 28 week extension period, in total 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* Diet/exercise therapy with sulfonylurea (SU) for at least eight weeks
* HbA1c greater than or equal to 7.0% and less than 10.0%
* BMI less than 35 kg/m2

Exclusion Criteria:

* Treatment with insulin within the last 12 weeks
* Treatment with any drug that could interfere with the glucose level
* Any serious medical condition
* Females who are pregnant, have intention of becoming pregnant or are breastfeeding

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Actual)
Dates: Start 2006-10; Primary Completion 2007-10 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Tokyo, Japan

REFERENCES:
- [Result] Seino Y, Rasmussen MF, Clauson P, Kaku K. The once-daily human glucagon-like peptide-1 analog, liraglutide, improves beta-cell function in Japanese patients with type 2 diabetes. J Diabetes Investig. 2012 Aug 20;3(4):388-95. doi: 10.1111/j.2040-1124.2012.00193.x. PMID 24843595
- [Result] Kaku K, Rasmussen MF, Clauson P, Seino Y. Improved glycaemic control with minimal hypoglycaemia and no weight change with the once-daily human glucagon-like peptide-1 analogue liraglutide as add-on to sulphonylurea in Japanese patients with type 2 diabetes. Diabetes Obes Metab. 2010 Apr;12(4):341-7. doi: 10.1111/j.1463-1326.2009.01194.x. PMID 20380655
- [Result] Alves C, Batel-Marques F, Macedo AF. A meta-analysis of serious adverse events reported with exenatide and liraglutide: acute pancreatitis and cancer. Diabetes Res Clin Pract. 2012 Nov;98(2):271-84. doi: 10.1016/j.diabres.2012.09.008. Epub 2012 Sep 23. PMID 23010561
- [Result] Jensen TM, Saha K, Steinberg WM. Is there a link between liraglutide and pancreatitis? A post hoc review of pooled and patient-level data from completed liraglutide type 2 diabetes clinical trials. Diabetes Care. 2015 Jun;38(6):1058-66. doi: 10.2337/dc13-1210. Epub 2014 Dec 12. PMID 25504028
- [Derived] Buse JB, Garber A, Rosenstock J, Schmidt WE, Brett JH, Videbaek N, Holst J, Nauck M. Liraglutide treatment is associated with a low frequency and magnitude of antibody formation with no apparent impact on glycemic response or increased frequency of adverse events: results from the Liraglutide Effect and Action in Diabetes (LEAD) trials. J Clin Endocrinol Metab. 2011 Jun;96(6):1695-702. doi: 10.1210/jc.2010-2822. Epub 2011 Mar 30. PMID 21450987
- [Derived] Hegedus L, Moses AC, Zdravkovic M, Le Thi T, Daniels GH. GLP-1 and calcitonin concentration in humans: lack of evidence of calcitonin release from sequential screening in over 5000 subjects with type 2 diabetes or nondiabetic obese subjects treated with the human GLP-1 analog, liraglutide. J Clin Endocrinol Metab. 2011 Mar;96(3):853-60. doi: 10.1210/jc.2010-2318. Epub 2011 Jan 5. PMID 21209033
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 49 sites in Japan
Pre-assignment Details: Subjects included were patients with type 2 diabetes treated with diet therapy and one sulphonylurea (SU) agent (glibenclamide, gliclazide or glimepiride). Subjects continued their current SU therapy with, as a rule, no change in the dose and dosage in the study. A total of 267 subjects were randomised, 3 subjects were not exposed to study drug.
Groups:
- 0.6 mg + SU: Liraglutide 0.6 mg/day in addition to subject's own sulphonylurea (glibenclamide, gliclazide or glimepiride) treatment
- 0.9 mg + SU: Liraglutide 0.9 mg/day in addition to subject's own sulphonylurea (glibenclamide, gliclazide or glimepiride) treatment
- SU Mono: Liraglutide placebo (0.6 mg/day or 0.9 mg/day) in addition to subject's own sulphonylurea (glibenclamide, gliclazide or glimepiride) treatment
Period: Overall Study
Arm/Group | 0.6 mg + SU | 0.9 mg + SU | SU Mono
Started | 88 (Exposed to study drug) | 88 (Exposed to study drug) | 88 (Exposed to study drug)
Completed | 78 (Completed 52 weeks treatment) | 84 (Completed 52 weeks treatment) | 66 (Completed 52 weeks treatment)
Not Completed | 10 | 4 | 22
Not completed — Adverse Event | 5 | 2 | 2
Not completed — Protocol Violation | 0 | 1 | 0
Not completed — Lack of Efficacy | 2 | 0 | 17
Not completed — Hypoglycaemia | 2 | 1 | 0
Not completed — Subject decision | 0 | 0 | 1
Not completed — Withdrawal of consent | 0 | 0 | 1
Not completed — Difficultulty in use of device | 0 | 0 | 1
Not completed — Unable to visit site on schedule | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 0.6 mg + SU | 0.9 mg + SU | SU Mono | Total
Number analyzed (Participants) | 88 | 88 | 88 | 264
Age, Customized [Number; unit: participants]
  20-29 | 0 | 1 | 0 | 1
  30-39 | 2 | 4 | 0 | 6
  40-49 | 16 | 5 | 19 | 40
  50-59 | 24 | 27 | 28 | 79
  60-69 | 30 | 32 | 30 | 92
  70- | 16 | 19 | 11 | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.1 (10.3) | 61.3 (11.0) | 58.6 (9.7) | 59.7 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 29 | 31 | 95
  Male | 53 | 59 | 57 | 169
BMI [Mean (Standard Deviation); unit: kg/m2] — Body Mass Index
  kg/m2 | 25.25 (3.58) | 24.40 (3.37) | 24.94 (3.96) | 24.86 (3.65)
Body weight [Mean (Standard Deviation); unit: kg] | 66.19 (12.03) | 64.53 (11.95) | 66.79 (13.66) | 65.84 (12.56)
Duration of diabetes [Mean (Standard Deviation); unit: years] — Number of years since diagnosis of diabetes
  years | 9.33 (5.77) | 11.61 (7.68) | 10.06 (7.28) | 10.33 (7.00)
HbA1c [Mean (Standard Deviation); unit: percentage of total haemoglobin] — Glycosylated Haemoglobin
  percentage of total haemoglobin | 8.48 (0.73) | 8.26 (0.71) | 8.44 (0.83) | 8.39 (0.76)

OUTCOME MEASURES:

1. Primary Outcome: Glycosylated Haemoglobin A1c (HbA1c) After 24 Weeks of Treatment
Time Frame: after 24 weeks of treatment
Population: Full Analysis Set (FAS) using LOCF (Last Observation Carried Forward) is all subjects who received at least one dose of study drug and have valid measurements both at baseline and at least one time point after baseline.
Measure: Least Squares Mean (Standard Error); unit: percentage of total haemoglobin
Arm/Group | 0.6 mg + SU | 0.9 mg + SU | SU Mono
Number analyzed (Participants) | 86 | 87 | 88
percentage of total haemoglobin | 7.02 (0.10) | 6.75 (0.11) | 8.02 (0.10)
Statistical Analysis 1: Comparison: 0.9 mg + SU vs SU Mono; ANOVA model included treatment group and pre-trial SU as fixed effects and HbA1C at baseline as a covariate. Two null hypotheses were statistically tested: H10: μ0.9 = μSU, H11: μ0.9 ≠ μSU H20: μ0.6 = μSU, H21: μ0.6 ≠ μSU where μ0.6, μ0.9 and μSU are population mean after 24-week treatment for 0.6 mg+SU, 0.9 mg+SU and SU mono, respectively. When the test of comparison between 0.9 mg+SU and SU mono was significant, the test of comparison between 0.6 mg+SU and SU mono was performed; Test type: Superiority or Other; p < 0.0001, ANOVA — A significance level of a two-sided 5% was used for statistical hypothesis testing; Least Squares Mean = -1.27, 95% CI [-1.51 to 1.02]
Statistical Analysis 2: Comparison: 0.6 mg + SU vs SU Mono; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANOVA; A significance level of a two-sided 5% was used for statistical hypothesis testing; Least Squares Mean = -1.00, 95% CI [-1.24 to -0.75]

2. Secondary Outcome: Glycosylated Haemoglobin A1c (HbA1c) After 52 Weeks of Treatment
Time Frame: after 52 weeks of treatment
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage of total haemoglobin
Arm/Group | 0.6 mg + SU | 0.9 mg + SU | SU Mono
Number analyzed (Participants) | 86 | 87 | 88
percentage of total haemoglobin | 7.42 (0.12) | 7.06 (0.13) | 8.39 (0.12)
Statistical Analysis 1: Comparison: 0.9 mg + SU vs SU Mono; 95% confidence interval for the mean difference (each liraglutide - SU monotherapy) was calculated under an analysis of variance (ANOVA) model with treatment group and pre-trial SU as fixed effects and corresponding baseline value as a covariate, and no statistical testing was performed; Test type: Superiority or Other; ANOVA; Least Squares Mean = -1.33, 95% CI [-1.62 to -1.04]
Statistical Analysis 2: Comparison: 0.6 mg + SU vs SU Mono; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; ANOVA; Least Squares Mean = -0.96, 95% CI [-1.25 to -0.67]

3. Secondary Outcome: Fasting Plasma Glucose After 24 Weeks of Treatment
Time Frame: after 24 weeks of treatment
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | 0.6 mg + SU | 0.9 mg + SU | SU Mono
Number analyzed (Participants) | 85 | 86 | 87
mg/dL | 132.2 (3.5) | 126.2 (3.5) | 158.8 (3.5)
Statistical Analysis 1: Comparison: 0.9 mg + SU vs SU Mono; ANOVA model included treatment group and pre-trial SU as fixed effects and corresponding baseline value as a covariate. Two null hypotheses were statistically tested, when the hypothesis μ0.9 = μ0.6 = μSU was rejected at a significance level of 5%: H10: μ0.9 = μSU, H11: μ0.9 ≠ μSU H20: μ0.6 = μSU, H21: μ0.6 ≠ μSU where μ0.6, μ0.9 and μSU are population mean after 24-week treatment for 0.6 mg+SU, 0.9 mg+SU and SU mono, respectively; Test type: Superiority or Other; p < 0.0001, ANOVA — To perform the pairwise comparisons simultaneously, a closed testing procedure was applied. When the hypothesis μ0.9 = μ0.6 = μSU was rejected, the 2 hypotheses of pairwise comparison were tested simultaneously both at significance level of 5%; Least Squares Mean = -32.4, 95% CI [-40.5 to -24.2]
Statistical Analysis 2: Comparison: 0.6 mg + SU vs SU Mono; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANOVA — [p-value comment as in outcome 3, analysis 1]; Least Squares Mean = -26.4, 95% CI [-34.5 to -18.2]

4. Secondary Outcome: Fasting Plasma Glucose After 52 Weeks of Treatment
Time Frame: after 52 weeks of treatment
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | 0.6 mg + SU | 0.9 mg + SU | SU Mono
Number analyzed (Participants) | 85 | 86 | 87
mg/dL | 140.3 (4.0) | 134.5 (4.1) | 164.6 (4.0)
Statistical Analysis 1: Comparison: 0.9 mg + SU vs SU Mono; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; ANOVA; Least Squares Mean = -30.2, 95% CI [-39.6 to -20.7]
Statistical Analysis 2: Comparison: 0.6 mg + SU vs SU Mono; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; ANOVA; Least Squares Mean = -24.4, 95% CI [-33.8 to -14.9]

5. Secondary Outcome: Postprandial Glucose AUC After 24 Weeks of Treatment
Description: Postprandial glucose AUC measured 0-3 hours after a meal after 24 weeks of treatment
Time Frame: after 24 weeks of treatment
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL *h
Arm/Group | 0.6 mg + SU | 0.9 mg + SU | SU Mono
Number analyzed (Participants) | 83 | 84 | 71
mg/dL *h | 614.58 (14.75) | 575.50 (15.01) | 725.72 (15.71)
Statistical Analysis 1: Comparison: 0.9 mg + SU vs SU Mono; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANOVA — [p-value comment as in outcome 3, analysis 1]; Least Squares Mean = -150.22, 95% CI [-186.32 to -114.12]
Statistical Analysis 2: Comparison: 0.6 mg + SU vs SU Mono; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANOVA — [p-value comment as in outcome 3, analysis 1]; Least Squares Mean = -111.15, 95% CI [-147.61 to -74.68]

6. Secondary Outcome: Postprandial Glucose AUC After 52 Weeks of Treatment
Description: Postprandial Glucose AUC measured 0-3 hours after a meal after 52 weeks of treatment
Time Frame: after 52 weeks of treatment
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL *h
Arm/Group | 0.6 mg + SU | 0.9 mg + SU | SU Mono
Number analyzed (Participants) | 78 | 83 | 68
mg/dL *h | 648.87 (16.09) | 589.98 (16.17) | 717.55 (17.08)
Statistical Analysis 1: Comparison: 0.9 mg + SU vs SU Mono; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; ANOVA; Least Squares Mean = -127.57, 95% CI [-166.91 to -88.24]
Statistical Analysis 2: Comparison: 0.6 mg + SU vs SU Mono; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; ANOVA; Least Squares Mean = -68.68, 95% CI [-108.91 to -28.45]

7. Secondary Outcome: Mean PG in 7-point Plasma Glucose Profile After 24 Weeks of Treatment
Description: Plasma glucose (PG) profile measured after 24 weeks of treatment. The 7 time points during the day were: Before breakfast, 120 minutes after start of breakfast, before lunch, 120 minutes after start of lunch, before dinner, 120 minutes after start of dinner, and at bedtime.
Time Frame: after 24 weeks of treatment
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | 0.6 mg + SU | 0.9 mg + SU | SU Mono
Number analyzed (Participants) | 80 | 82 | 80
mg/dL | 160.20 (4.44) | 150.05 (4.56) | 194.50 (4.61)
Statistical Analysis 1: Comparison: 0.9 mg + SU vs SU Mono; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANOVA — [p-value comment as in outcome 3, analysis 1]; Least Squares Mean = -44.45, 95% CI [-55.02 to -33.89]
Statistical Analysis 2: Comparison: 0.6 mg + SU vs SU Mono; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANOVA — [p-value comment as in outcome 3, analysis 1]; Least Squares Mean = -34.30, 95% CI [-45.06 to -23.54]

8. Secondary Outcome: Mean PG in 7-point Plasma Glucose Profile After 52 Weeks of Treatment
Description: 7-point plasma glucose (PG) profile measured after 52 weeks of treatment. The 7 time points during the day were: Before breakfast, 120 minutes after start of breakfast, before lunch, 120 minutes after start of lunch, before dinner, 120 minutes after start of dinner, and at bedtime.
Time Frame: after 52 weeks of treatment
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | 0.6 mg + SU | 0.9 mg + SU | SU Mono
Number analyzed (Participants) | 81 | 80 | 82
mg/dL | 171.42 (5.11) | 159.58 (5.30) | 205.92 (5.25)
Statistical Analysis 1: Comparison: 0.6 mg + SU vs SU Mono; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; ANOVA; Least Squares Mean = -34.49, 95% CI [-46.77 to -22.22]
Statistical Analysis 2: Comparison: 0.9 mg + SU vs SU Mono; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; ANOVA; Least Squares Mean = -46.34, 95% CI [-58.49 to -34.18]

9. Secondary Outcome: Mean Postprandial PG Increment in 7-point Plasma Glucose Profile After 24 Weeks of Treatment
Description: Mean postprandial plasma glucose (PG) increment in 7-point plasma glucose profile, ie the mean of the difference of plasma glucose measured before and after a meal, after 24 weeks of treatment. The 7 time points during the day were: Before breakfast, 120 minutes after start of breakfast, before lunch, 120 minutes after start of lunch, before dinner, 120 minutes after start of dinner, and at bedtime.
Time Frame: after 24 weeks of treatment
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | 0.6 mg + SU | 0.9 mg + SU | SU Mono
Number analyzed (Participants) | 81 | 82 | 82
mg/dL | 86.38 (4.65) | 68.34 (4.78) | 79.71 (4.75)
Statistical Analysis 1: Comparison: 0.9 mg + SU vs SU Mono; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.0433, ANOVA — [p-value comment as in outcome 3, analysis 1]; Least Squares Mean = -11.37, 95% CI [-22.40 to -0.34]
Statistical Analysis 2: Comparison: 0.6 mg + SU vs SU Mono; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.2359, ANOVA — [p-value comment as in outcome 3, analysis 1]; Least Squares Mean = 6.67, 95% CI [-4.39 to 17.73]

10. Secondary Outcome: Mean Postprandial PG Increment in 7-point Plasma Glucose Profile After 52 Weeks of Treatment
Description: Mean postprandial plasma glucose (PG) increment in 7-point plasma glucose profile, ie the mean of the difference of plasma glucose measured before and after a meal, after 52 weeks of treatment. The 7 time points during the day were: Before breakfast, 120 minutes after start of breakfast, before lunch, 120 minutes after start of lunch, before dinner, 120 minutes after start of dinner, and at bedtime.
Time Frame: after 52 weeks of treatment
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | 0.6 mg + SU | 0.9 mg + SU | SU Mono
Number analyzed (Participants) | 82 | 80 | 85
mg/dL | 82.28 (4.81) | 76.09 (5.00) | 89.39 (4.86)
Statistical Analysis 1: Comparison: 0.9 mg + SU vs SU Mono; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; ANOVA; Least Squares Mean = -13.30, 95% CI [-24.69 to -1.90]
Statistical Analysis 2: Comparison: 0.6 mg + SU vs SU Mono; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; ANOVA; Least Squares Mean = -7.11, 95% CI [-18.42 to 4.21]

11. Secondary Outcome: Body Weight After 24 Weeks of Treatment
Time Frame: after 24 weeks of treatment
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | 0.6 mg + SU | 0.9 mg + SU | SU Mono
Number analyzed (Participants) | 87 | 87 | 88
kg | 65.77 (0.23) | 65.34 (0.24) | 64.59 (0.23)
Statistical Analysis 1: Comparison: 0.9 mg + SU vs SU Mono; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.0071, ANOVA — [p-value comment as in outcome 3, analysis 1]; Least Squares Mean = 0.75, 95% CI [0.21 to 1.30]
Statistical Analysis 2: Comparison: 0.6 mg + SU vs SU Mono; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANOVA — [p-value comment as in outcome 3, analysis 1]; Least Squares Mean = 1.18, 95% CI [0.63 to 1.73]

12. Secondary Outcome: Body Weight After 52 Weeks of Treatment
Time Frame: after 52 weeks of treatment
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | 0.6 mg + SU | 0.9 mg + SU | SU Mono
Number analyzed (Participants) | 87 | 87 | 88
kg | 65.96 (0.26) | 65.87 (0.27) | 64.83 (0.26)
Statistical Analysis 1: Comparison: 0.9 mg + SU vs SU Mono; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; ANOVA; Least Squares Mean = 1.04, 95% CI [0.42 to 1.66]
Statistical Analysis 2: Comparison: 0.6 mg + SU vs SU Mono; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; ANOVA; Least Squares Mean = 1.13, 95% CI [0.51 to 1.75]

13. Secondary Outcome: Hypoglycaemic Episodes
Description: Hypoglycaemic episodes measured over 52 weeks of treatment. Hypoglycaemic episodes were defined as major, minor, or symptoms only. Major if the subject was unable to treat her/himself. Minor if subject was able to treat her/himself and plasma glucose was below 3.1 mmol/L. Symptoms only if subject was able to treat her/himself and with no plasma glucose measurement or plasma glucose higher than or equal to 3.1 mmol/L.
Time Frame: over 52 weeks of treatment
Population: Full Analysis Set (FAS) consists of all subjects who received at least one dose of study drug.
Measure: Number; unit: number of events per year of exposure
Arm/Group | 0.6 mg + SU | 0.9 mg + SU | SU Mono
Number analyzed (Participants) | 88 | 88 | 88
number of events per year of exposure
  All hypoglycaemic episodes | 3.131 | 3.715 | 2.990
  Major | 0.0000 | 0.0000 | 0.0000
  Minor | 1.438 | 1.365 | 1.285
  Symptoms only | 1.693 | 2.350 | 1.705
Statistical Analysis 1: Comparison: 0.9 mg + SU vs SU Mono; The relative risk for 'All hypoglycaemic episodes' and 95% confidence interval are based on a generalised linear negative-binomial model, which included treatment group as a fixed effect and log of exposure time as an offset variable; Test type: Superiority or Other; Negative binomial regression; Rate ratio = 1.59, 95% CI [0.86 to 2.96]
Statistical Analysis 2: Comparison: 0.9 mg + SU vs SU Mono; The relative risk for 'Minor episodes' and 95% confidence interval are based on a generalised linear negative-binomial model, which included treatment group as a fixed effect and log of exposure time as an offset variable; Test type: Superiority or Other; Negative binomial regression model; Rate ratio = 1.18, 95% CI [0.56 to 2.47]
Statistical Analysis 3: Comparison: 0.9 mg + SU vs SU Mono; The relative risk for 'Symptoms only' and 95% confidence interval are based on a generalised linear negative-binomial model, which included treatment group as a fixed effect and log of exposure time as an offset variable; Test type: Superiority or Other; Negative binomial regression model; Rate ratio = 1.80, 95% CI [0.92 to 3.54]
Statistical Analysis 4: Comparison: 0.6 mg + SU vs SU Mono; [analysis description as in outcome 13, analysis 1]; Test type: Superiority or Other; Negative binomial regression model; Rate ratio = 1.62, 95% CI [0.85 to 3.07]
Statistical Analysis 5: Comparison: 0.6 mg + SU vs SU Mono; [analysis description as in outcome 13, analysis 2]; Test type: Superiority or Other; Negative binomial regression model; Rate ratio = 1.48, 95% CI [0.69 to 3.17]
Statistical Analysis 6: Comparison: 0.6 mg + SU vs SU Mono; The relative risk for 'Symptoms only episodes' and 95% confidence interval are based on a generalised linear negative-binomial model, which included treatment group as a fixed effect and log of exposure time as an offset variable; Test type: Superiority or Other; Negative binomial regression model; Rate ratio = 1.45, 95% CI [0.72 to 2.91]

ADVERSE EVENTS:
Time Frame: Adverse events were collected in a time span over 52 weeks.
Description: The safety analysis population consists of all subjects exposed to study drug (Full Analysis Set, FAS).
Arm/Group | 0.6 mg + SU | 0.9 mg + SU | SU Mono
Serious Adverse Events (participants affected / at risk) | 4/88 | 3/88 | 5/88
Other Adverse Events (participants affected / at risk) | 68/88 | 68/88 | 59/88
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0.6 mg + SU (N=88) | 0.9 mg + SU (N=88) | SU Mono (N=88)
Sudden hearing loss (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Colitis ischaemic (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Bursitis infective (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Benign neoplasm of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Epiglottic cyst (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Cataract operation (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0.6 mg + SU (N=88) | 0.9 mg + SU (N=88) | SU Mono (N=88)
Nasopharyngitis (Infections and infestations) | 37 (63) | 38 (51) | 35 (61)
Diarrhoea (Gastrointestinal disorders) | 7 (8) | 14 (17) | 7 (10)
Constipation (Gastrointestinal disorders) | 8 (9) | 11 (12) | 4 (7)
Dental caries (Gastrointestinal disorders) | 5 (5) | 5 (5) | 1 (1)
Gastritis (Gastrointestinal disorders) | 3 (3) | 4 (4) | 8 (8)
Back pain (Musculoskeletal and connective tissue disorders) | 10 (10) | 7 (8) | 6 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (6) | 3 (3) | 1 (1)
Diabetic retinopathy (Eye disorders) | 8 (8) | 11 (11) | 7 (7)
Dizziness (Nervous system disorders) | 5 (7) | 6 (7) | 2 (2)
Headache (Nervous system disorders) | 10 (11) | 4 (4) | 8 (9)
Hypoaesthesia (Nervous system disorders) | 5 (6) | 0 (0) | 5 (5)
Alanine aminotransferase increased (Investigations) | 6 (7) | 2 (2) | 1 (1)
Malaise (General disorders) | 5 (6) | 1 (2) | 5 (6)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 9 (12) | 6 (8) | 5 (5)
Fall (Injury, poisoning and procedural complications) | 5 (5) | 2 (3) | 2 (2)
Hypertension (Vascular disorders) | 5 (5) | 3 (3) | 4 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Novo Nordisk acknowledges the Investigator's right to publish the entire results of the trial. Any such scientific paper, presentation, communication or other information concerning the investigation described in this protocol, must be submitted in writing to Novo Nordisk Trial Manager prior to submission for publication/presentation for comments. Comments will be given within four weeks from receipt of the manuscript.